CLINICAL TRIAL: NCT05509777
Title: A Phase 3, Multicenter, Randomized Clinical Study to Evaluate Mirikizumab in Pediatric Crohn's Disease
Brief Title: A Study of Mirikizumab (LY3074828) in Pediatric Participants With Crohn's Disease
Acronym: AMAY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16632; I6T-MC-AMAY (Other: Eli Lilly and Company); MACARONI-23 (Other: Eli Lilly and Company); PLATFORMPBCRD3001 (Other: Eli Lilly and Company); I6T-MC-PIBD (Other: Eli Lilly and Company); 2024-511472-32-00 (EU CTIS Number)
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Crohn's Disease
Keywords: Inflammatory Bowel Disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — mirikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Mirikizumab Dose 1 (Experimental): Mirikizumab administered intravenously (IV) or subcutaneously (SC) in participants that weigh greater than (>) 40 kilograms (kg).
  Interventions: Drug: Mirikizumab
- Mirikizumab Dose 2 (Experimental): Mirikizumab administered IV or SC in participants that weigh >20 kg to less than or equal to (≤) 40 kg.
  Dosing is based on assessments of the participant's weight and appropriate weight class.
  Interventions: Drug: Mirikizumab
- Mirikizumab Dose 3 (Experimental): Mirikizumab administered IV or SC in participants that weigh greater than or equal to (≥) 9 kg to less than or equal to ≤20 kg.
  Dosing is based on assessments of the participant's weight and appropriate weight class.
  Interventions: Drug: Mirikizumab

INTERVENTIONS:
Drug: Mirikizumab — Administered IV or SC
  Other Names: LY3074828

SUMMARY:
Study participants will be screened during the platform study and randomly assigned to receive mirikizumab or another intervention. The purpose of the mirikizumab study is to evaluate efficacy, safety, tolerability, and how well mirikizumab absorbs into the body of pediatric participants with Crohn's disease.

Study periods for the intervention-specific appendix (ISA) will be as follows:

* A 12-week induction period
* A maintenance period from Week 12 to Week 52, and
* A safety follow-up period up to 16 weeks.

The study will last about 74 weeks and may include up to 19 visits.

DETAILED DESCRIPTION:
Participants screened in the MACARONI-23 Platform study could be randomized to mirikizumab to participate in this intervention specific arm of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of CD or fistulizing CD, with active colitis, ileitis, or ileocolitis, confirmed at any time in the past by clinical, endoscopic, and histologic criteria.
* Participants have moderately to severely active CD (as defined by a baseline PCDAI score ≥30).
* Participants must have endoscopy with evidence of active CD defined as SES-CD score ≥6 (or ≥4 for participants with isolated ileal disease) within 1 month of receiving study intervention at Week 0.
* Participants must have a documented history of inadequate response, loss of response or intolerance to at least one medication used to treat CD, which may include immunomodulators, oral or IV corticosteroids, a biologic therapy or a JAK inhibitor.

Exclusion Criteria:

* Participants must not have complications of CD such as symptomatic strictures or stenosis, short gut syndrome, or any other manifestations that might be anticipated to require surgery.
* Participants must not have an abscess.
* Participants must not have any kind of bowel resection within 26 weeks or any other intra-abdominal surgery within 12 weeks of baseline.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Clinical Response by Pediatric Crohn's Disease Activity Index (PCDAI) at Week 12 and Endoscopic Response by Simple Endoscopic Score for CD (SES-CD) at Week 52 | Baseline to Week 52
  Clinical response based on PCDAI, and endoscopic response based on SES-CD.
Percentage of Participants with a Clinical Response by PCDAI at Week 12 and Clinical Remission by PCDAI at Week 52 | Baseline to Week 52
  Clinical response based on PCDAI, and clinical remission based on PCDAI.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Clinical Response by PCDAI | Week 12
  Clinical response based on PCDAI.
Percentage of Participants Achieving Clinical Response by Clinical Disease Activity Index (CDAI) | Week 12
  Clinical response based on CDAI for participants ≥12 years of age
Percentage of Participants Achieving Clinical Remission by PCDAI | Week 12
  Clinical remission based on PCDAI.
Percentage of Participants Achieving Clinical Remission by CDAI | Week 12
  Clinical remission based on CDAI for participants ≥12 years of age.
Percentage of Participants Who Achieve PCDAI Clinical Response at Week 12 and PCDAI Clinical Remission and Endoscopic Remission at Week 52 | Baseline to Week 52
Percentage of Participants Who Achieve PCDAI Clinical Remission and Endoscopic Remission at Week 52 | Week 52
Percentage of Participants Achieving Clinical Response by PCDAI at Week 12 and Endoscopic Remission by SES-CD at Week 52 | Baseline to Week 52
Change from Baseline in C-reactive Protein (CRP) | Baseline, Week 12
Change from Baseline in CRP | Baseline, Week 52
Change from Baseline in Fecal calprotectin | Baseline, Week 12
Change from Baseline in Fecal calprotectin | Baseline, Week 52
Percentage of Participants Achieving Clinical Response PCDAI at Week 12 and Clinical Remission by CDAI at Week 52 | Baseline to Week 52
  Clinical response by PCDAI, CDAI for participants ≥12 years of age
Percentage of Participants Achieving Endoscopic Response | Week 52
Percentage of Participants Achieving Clinical Remission by PCDAI | Week 52
  Clinical remission based on PCDAI
Percentage of Participants Achieving Clinical Response by PCDAI at Week 12 and PCDAI Clinical Remission without the use of Corticosteroids and Who Did Not Have Crohn's Disease (CD)-Related Surgery at Week 52 | Baseline to Week 52
  Clinical response and clinical remission by PCDAI
Pharmacokinetics (PK): Clearance of Mirikizumab | Baseline through Week 52
Pharmacokinetics (PK): Volume of Distribution of Mirikizumab | Baseline through Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (85):
- United States (16):
  - University of California San Diego, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Emory University, Atlanta, Georgia
  - Children's Center for Digestive Health Care, LLC, Atlanta, Georgia
  - Riley Childrens Hospital, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Atlantic Children's Health--Pediatric Gastroenterology, Morristown, New Jersey
  - Weill Cornell Medical College (WCMC) - Judith Jaffe Multiple Sclerosis Center (JJMSC), New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center/New York Presbyterian, New York, New York
  - Childrens Medical Center, Dayton, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Children's Medical Center, Fort Worth, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Seattle Children's Hospital, Seattle, Washington
- AKH - Medizinische Universtität Wien, Vienna, Austria
- Belgium (4):
  - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
- Brazil (7):
  - Hospital PUC-CAMPINAS, Campinas
  - Hospital Pequeno Príncipe, Curitiba-PR
  - Hospital das Clínicas - UFG (Universidade Federal de Goiás), Goiânia
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - NDI - Nucleo de Doenças Infecciosas, Santos Dumont
  - Integral Pesquisa e Ensino, Votuporanga
- Canada (4):
  - IWK Health Centre, Halifax
  - London Health Sciences Centre (LHSC) - Victoria Hospital, London
  - The Hospital for Sick Children, Toronto
  - Children's & Women's Health Centre of British Columbia, Vancouver
- URC CIC, Paris, France
- Israel (6):
  - Soroka Medical Center, Beersheba
  - Shamir Medical Center (Assaf Harofeh), Israel
  - Shaare Zedek, Jerusalem
  - Hadassah University Hospital, Ein Kerem,, Jerusalem
  - Schneider Children's Medical Center, Petah Tikva
  - Kaplan Medical Center, Pediatric Gastroenterology Dept., Rehovot
- Italy (6):
  - Asst Papa Giovanni Xxiii Bergamo, Bergamo
  - Azienda USL di Bologna, Bologna
  - SOC Gastroenterologia e Nutrizione - AOU Meyer (Primo Piano Ala OVEST, accettazione DH centralizzato), Florence
  - Ospedale dei Bambini Vittore Buzzi, Milan
  - Ospedale Pediatrico Bambino Gesù, Roma
  - Gastroenterologia ed epatologia pediatrica (Piano terra della Clinica Pediatrica), Roma
- Japan (12):
  - Juntendo University Hospital, Bunkyō City
  - Hirosaki University Hospital, Hirosaki
  - Kagoshima University Hospital, Kagoshima
  - Kokikai Tsujinaka Hospital Kashiwanoha, Kashiwa-shi
  - Kobe University Hospital, Kobe
  - Saga University Hospital, Saga
  - Miyagi Children's Hospital, Sendai
  - National Center for Child Health and Development, Setagaya-ku
  - Mie University Hospital, Tsu
  - Yamaguchi University Hospital, Ube
  - Saiseikai Yokohamashi Tobu Hospital, Yokohama
  - Yokohama City University Medical Center, Center of IBD, Yokohama
- Erasmus Medisch Centrum, Rotterdam, Netherlands
- Norway (4):
  - Akershus Universitetssykehus, Nordbyagen
  - Oslo University Hospital, Oslo
  - Universitetssykehuset Nord-Norge, Tromsø
  - St-Olavs Hospital, Trondheim
- Poland (5):
  - Uniwersytecki Szpital Dziecięcy w Krakowie, Krakow
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów
  - Centrum Zdrowia MDM, Warsaw
  - Warsaw IBD Point Profesor Kierkus, Warsaw
  - Instytut Pomnik-Centrum Zdrowia Dziecka, Warsaw
- Portugal (3):
  - Centro Clínico Académico - Braga (2CA-Braga) (Hospital de Braga), Braga
  - Centro Hospitalar de Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar de São João, E.P.E., Porto
- South Korea (5):
  - Inje University Haeundae Paik Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Spain (4):
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Sant Joan de Deu, Esplugues de Llobregat
  - Corporacio Sanitaria Parc Tauli, Sabadell
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (6):
  - Royal Hospital for Children and Young People, Edinburgh
  - Oxford University Hospitals NHS trust John Radcliffe hospital, Headington
  - Great Ormond Street Hospital For Children NHS Foundation Trust, London
  - Manchester University NHS Foundation Trust, Manchester
  - Sheffield Children's Hospital, Sheffield
  - Royal London Hospital, Whitechapel

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Mirikizumab (LY3074828) in Pediatric Participants With Crohn's Disease (AMAY) — https://trials.lilly.com/en-US/trial/356367